CLINICAL TRIAL: NCT06687161
Title: Neuromodulation and Cognitive Behavioral Therapy for Insomnia in MCI
Brief Title: Treating Insomnia in Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Principal Investigator, Peter J. Fried, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000708; A2024034S (Other Grant/Funding Number: BrightFocus Foundation)
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment (MCI); Insomnia
Keywords: transcranial magnetic stimulation; neuromodulation; cognitive behavioral therapy; CBT-I; TMS; sleep
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders | interventions — Transcranial Magnetic Stimulation; Therapeutics; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study will test the combination of neuromodulation by repetitive transcranial magnetic stimulation (rTMS) with cognitive behavioral therapy for insomnia (CBT-I). All participants will receive the active intervention. Participants will be randomized to receive one or two treatments of rTMS per day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- One (1) TMS treatment per day plus CBT-I (Active Comparator): One (1) daily treatment of intermittent theta-burst stimulation (iTBS) applied to the left dorsolateral prefrontal cortex (L-DLPFC) for 10 days (2 weeks) followed by a 9-week Internet-delivered cognitive behavioral therapy for insomnia (CBT-I) program
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) therapy; Behavioral: Cognitive behavioral therapy for insomnia (CBT-I)
- Two (2) TMS treatments per day plus CBT-I (Active Comparator): Two (2) daily treatments, spaced 1 hour apart, of intermittent theta-burst stimulation (iTBS) applied to the left dorsolateral prefrontal cortex (L-DLPFC) for 10 days (2 weeks) followed by a 9-week Internet-delivered cognitive behavioral therapy for insomnia (CBT-I) program
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) therapy; Behavioral: Cognitive behavioral therapy for insomnia (CBT-I)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) therapy — Each treatment consists of 600 TMS pulses (~3 minutes) applied to the L-DLPFC
  Other Names: Intermittent theta-burst stimulation (iTBS)
Behavioral: Cognitive behavioral therapy for insomnia (CBT-I) — 9-week fully-automated, Internet-delivered CBT-I program: SHUTi OASIS (Sleep Healthy Using the Internet for Older Adult Sufferers of Insomnia and Sleeplessness)
  Other Names: SHUTi OASIS

SUMMARY:
The goal of this study is to test a new way to improve sleep quality in persons living with mild cognitive impairment. The treatment combines a safe and gentle way to stimulate the brain, called transcranial magnetic stimulation, with a psychological treatment, called cognitive behavioral therapy for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older
* Speak and read English
* Clinical diagnosis of MCI or Subjective Cognitive Impairment (SCI)-a perceived gradual worsening in cognitive ability relative to one's younger self, or peer group-reported by either the participant or informant
* Reported insomnia symptoms (sleep-onset and/or sleep maintenance) that cause significant distress or impairment in social, occupational, or other areas of functioning over the past three months
* Have access to an Internet-enabled computer or tablet at home, or ability to connect a BIDMC-provided tablet to the internet, with private space to complete cognitive testing
* Capable of and willing to provide written informed consent

Exclusion Criteria:

* Evidence of significant cognitive impairment or dementia
* Contraindications for TMS or MRI
* Current psychological treatment for insomnia
* Uncontrolled moderate-to-severe obstructive sleep apnea or other untreated sleep disorder (e.g., Restless Leg Syndrome, Periodic Limb Movement Disorder, parasomnia). Sleep apnea that is managed (e.g., regular use of a CPAP) and stable for ≥3 months is allowed.
* Diagnosis of Parkinson's disease, Huntington's disease, Lewy-Body disease, or other neurological condition known to impact sleep
* Current diagnosis of major psychiatric disorder (well-controlled depression or anxiety is permitted)
* Current opiate/opioid use
* Alcohol or drug abuse within the past year
* Irregular sleep schedule (bedtime before 8pm/after 2am OR wake time before 4am/after 10am), unless participant states they are willing and able to change if prompted.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | Baseline, Week 3 (Post-TMS), Week 12 (Post-CBT-I), 6 months (follow-up)
  The Insomnia Severity Index (ISI) is a brief self-assessment tool used to measure the severity of insomnia. It consists of seven questions that evaluate sleep problems, their impact on daily life, and the individual's level of concern about their sleep issues. The total score helps to categorize the severity of insomnia from mild to severe.
Paired Associative Learning test (CANTAB) | Baseline, Week 3, Week 12, 6 Months
  The Paired Associative Learning (PAL) test is a computer-based cognitive assessment that evaluates memory and learning. In the test, participants are shown patterns and must remember the locations of these patterns on a screen. It is commonly used to assess spatial memory and detect early signs of memory-related conditions like Alzheimer's disease.
Spatial Working Memory test (CANTAB) | Baseline, Week 3, Week 12, 6 months
  The Spatial Working Memory (SWM) test is a computer-based task used to assess the ability to retain and manipulate spatial information. Participants must find hidden tokens within a series of boxes while avoiding revisiting previously searched locations. This test measures executive function and memory, and is often used in research on conditions affecting cognitive function.

SECONDARY OUTCOMES:
Multidimensional Fatigue Symptoms Inventory | Baseline, Week 3, Week 12, 6 months
  The Multidimensional Fatigue Symptom Inventory (MFSI) is a questionnaire designed to assess different aspects of fatigue. It measures five dimensions: general fatigue, emotional fatigue, physical fatigue, mental fatigue, and vigor (energy levels). The tool helps to provide a comprehensive understanding of an individual's fatigue symptoms and their impact on daily functioning.
Center for Epidemiologic Studies Depression scale | Baseline, Week 3, Week 12, 6 months
  The Center for Epidemiologic Studies Depression scale (CES-D) is a self-report questionnaire designed to measure symptoms of depression in the general population. It consists of 20 questions that assess mood, behavior, and physical symptoms associated with depression over the past week. The CES-D is commonly used in research and clinical settings to screen for depressive symptoms and monitor changes in mood.
Match to Sample Visual Search test (CANTAB) | Baseline, Week 3, Week 12, 6 months
  The Match to Sample Visual Search (MTS) test is a computerized assessment that measures visual recognition and attention. In the test, participants are shown a sample pattern and must quickly identify the matching pattern from a selection of similar images. It evaluates processing speed, visual memory, and attention to detail, and is often used to study cognitive functions in various neurological and psychiatric conditions.
Montreal Cognitive Assessment | Baseline, Week 3, Week 12, 6 months
  The Montreal Cognitive Assessment (MoCA) is a quick test used by doctors and other healthcare professionals to check a person's thinking and memory skills. It takes about 10-15 minutes and looks at things like attention, memory, language, and problem-solving. It's often used to help spot early signs of conditions like dementia or mild cognitive impairment.
Sleep efficiency (sleep diaries) | Week 3, Week 13, 6 months
  Sleep Efficiency is a measure derived from sleep diaries that indicates the percentage of time spent asleep while in bed, relative to the total time spent in bed. It is calculated by dividing the total sleep time by the total time in bed and multiplying by 100 to get a percentage. A higher sleep efficiency typically suggests more consolidated sleep, while lower sleep efficiency can indicate difficulties with sleep onset or frequent awakenings.
Sleep After Wake Onset (sleep diaries) | Week 3, Week 13, Week 40
  Sleep After Wake Onset (SAWO) is a measure derived from sleep diaries that captures the amount of time a person manages to sleep after experiencing an initial awakening during the night. It represents the total time spent asleep between waking up and the final morning awakening, providing insight into the continuity of sleep and the ability to return to sleep after disruptions.
Sleep Onset Latency (sleep diaries) | Week 3, Week 13, Week 40
  Sleep Onset Latency (SOL) is a measure derived from sleep diaries that indicates the amount of time it takes to fall asleep after going to bed with the intention of sleeping. It is typically recorded in minutes and reflects how easily a person initiates sleep. Longer sleep onset latency may indicate difficulty falling asleep, while shorter latency suggests quicker sleep initiation.
Sleep efficiency (actigraphy) | Week 3, Week 13, 6 months
  Sleep Efficiency is a measure derived from actigraphy that indicates the percentage of time spent asleep while in bed, relative to the total time spent in bed. It is calculated by dividing the total sleep time by the total time in bed and multiplying by 100 to get a percentage. A higher sleep efficiency typically suggests more consolidated sleep, while lower sleep efficiency can indicate difficulties with sleep onset or frequent awakenings.
Sleep After Wake Onset (actigraphy) | Week 3, Week 13, Week 40
  Sleep After Wake Onset (SAWO) is a measure derived from actigraphy that captures the amount of time a person manages to sleep after experiencing an initial awakening during the night. It represents the total time spent asleep between waking up and the final morning awakening, providing insight into the continuity of sleep and the ability to return to sleep after disruptions.
Sleep Onset Latency (actigraphy) | Week 3, Week 13, Week 40
  Sleep Onset Latency (SOL) is a measure derived from actigraphy that indicates the amount of time it takes to fall asleep after going to bed with the intention of sleeping. It is typically recorded in minutes and reflects how easily a person initiates sleep. Longer sleep onset latency may indicate difficulty falling asleep, while shorter latency suggests quicker sleep initiation.

OTHER OUTCOMES:
Cortical Plasticity | Baseline (first day of TMS therapy)
  Cortical plasticity is a measure of the efficacy of long-term potentiation (LTP)-neuroplasticity. It will be measured as the change in the TMS-evoked EEG potential (TEP) following iTBS.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available for qualified researchers approximately.
Supporting Information: Study Protocol
Time Frame: Approximately 1 year following the conclusion of the study for at least 5 years
Access Criteria: Researchers at universities and academic medical centers can request de-identified data by sending an email to the PI and describing the nature of the request.